CLINICAL TRIAL: NCT04435548
Title: Multi-Omic Microbiome Study: Characterization of the Human Microbiota Among Chinese Population to Understant How the Microbiome Impacts Human Health.
Brief Title: Westlake Gut Microbiome Study
Status: Withdrawn | Type: Observational
Why Stopped: Owing to the impact of COVID-19, the study had to be withdrawn.
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20190901ZJS0011
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood, saliva, urine and feces.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Westlake Gut Microbiome study is a prospective cohort study. This project aims to characterize the gut microbiome among Chinese populations from different regions of China, and explore the relationships between gut microbiota and human health. Human fecal samples will be collected from the participants and muli-omics detection and analysis will be performed.

DETAILED DESCRIPTION:
In the first phase of the study (also a pilot study), the investigators will create a longitudinal datasets from a students-based cohort in Westlake University. Information about demography, life style, diet, medical history, physical activity will be recorded, clinical examinations such as blood glucose, body composition and electroencephalogram will be examined, and biological samples including blood, saliva, urine and feces, will be collected.

In the second phase, the investigators will expand to include eligible participants from at least 10 provinces of China, which are located at different regions. Similar to the procedures in phase 1 stage, information about demography, life style, diet, medical history, physical activity will be recorded, clinical examinations will be performed, and biological samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

Participants or her/his legal guardian are able to report the antibiotics use during the past 3 months; Participants or her/his legal guardian are able to understand and respond to the online questionairs; Participants or her/his legal guardian are able and willing to collect the biological samples as instructed; Participants or her/his legal guardian are able and willing to provide written informed consent; -

Exclusion Criteria:

Those with serious fundamental diseases or infectious diseases; and those with other conditions that not suitable to participate in this study, as considered by the investigators.

-

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the participants should be Chinese residents, regardless of the ethics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | 36 months
  Fecal microbiome will be analyzed by 16S rRNA gene sequencing and metagenome sequencing.
Metabolomics of serum and gut microbiome | 36 months
  Metabolomics of serum and gut microbiome will be analyzed by liquid chromatograph-mass spectrometer (LC/MS)
Proteomic profiling of serum | 36 months
  Proteomic characterization of serum will be analyzed by liquid chromatograph-mass spectrometer (LC/MS)

SECONDARY OUTCOMES:
Body composition | 36 months
  Body composition will be analyzed using composition automatic analyzer at the time point of sample collection by compostion automatic analyzer.
Biochemical examination of blood samples | 36 months
  Blood glucose, blood lipids, serum cytokines will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided